CLINICAL TRIAL: NCT01652807
Title: An 8-Week Hatha Yoga Intervention for Stress and Mental Health
Brief Title: Yoga for Stress and Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern Methodist University (Other)
Responsible Party: Principal Investigator, Jasper Smits, Ph.D., Associate Professor, Southern Methodist University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012-028-DEBL
Record Dates: First submitted 2012-07-23; First posted 2012-07-30 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Physiological Stress; Psychological Distress; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga (Experimental): The yoga intervention will last eight weeks and include two 90-minute sessions each week. Each yoga session will consist of the same series of 26 Hatha yoga postures, two breathing exercise, and two savasanas (i.e., a resting/relaxation posture), in a room heated to 104 degrees Fahrenheit, which aids in safe muscle stretching.
  Interventions: Behavioral: Hatha Yoga
- Waitlist (Delayed Yoga) (No Intervention): Participants assigned randomly to the control condition will provided an identical free two-month membership to Bikram Yoga Dallas after the week following their post-intervention session.

INTERVENTIONS:
Behavioral: Hatha Yoga — The yoga intervention will last eight weeks and include two 90-minute sessions each week. Each yoga session will consist of the same series of 26 Hatha yoga postures, two breathing exercise, and two savasanas (i.e., a resting/relaxation posture), in a room heated to 104 degrees Fahrenheit, which aids in safe muscle stretching. Each participant will be given a yoga studio scan card valid for two months, and, like all yoga studio members, they will be required to scan their card prior to their yoga class.
  Arms: Yoga

SUMMARY:
This study looks at an 8-week hatha yoga intervention for women reporting high levels of stress, a risk factor for various forms of psychopathology.

DETAILED DESCRIPTION:
Yoga practice appears to reduce stress and associated emotions. Specifically, yoga has been associated with significant decreases in depression, anxiety, and perceived stress. These findings underscore the promise of yoga practice for improving mental health in women prone to stress.

This study aims to examine the feasibility, acceptability, and efficacy of an eight-week Hatha Yoga intervention for improving stress and mental health. To this end, the investigators will recruit 40 women high in stress to receive an 8-week hatha yoga intervention consisting of two weekly 90-minute sessions. At baseline and at post-intervention, participants will undergo several cognitive, emotional, and behavioral assessments, followed by a relaxation time. Primary feasibility outcomes will be the time required to recruit 40 participants, the number of screen failures, participant retention and participant adherence to the study protocol. Acceptability will be evaluated with questionnaires and an interview during the final visit. Primary efficacy outcomes will be group differences in pre- to post-intervention change in perceived stress and various mental health parameters.

ELIGIBILITY:
Inclusion Criteria:

* Female patients between the ages of 25 and 45. We only will only include women in this age range due to age-related variations in estrogen levels that effect HPA reactivity in women (Seeman, Singer, Wilkinson & McEwen, 2001).
* Sedentary as defined by moderate-intensity exercise less than 60 minutes per week (this definition is consistent with that employed in previous studies of exercise interventions; e.g., Dunn et al., 2005; Trivedi et al., 2006). This criterion was selected in order to be able to test the effects of the yoga intervention.
* Written physician approval/medical clearance to participate in an exercise/yoga protocol.
* Capable and willing to give written informed consent, to understand inclusion and exclusion criteria.

Exclusion Criteria:

* Have practiced yoga or engaged in other mind-body practices (e.g., tai chi, meditation) regularly (i.e., once a week or more) within the last year.
* Lifetime history of psychotic disorders of any type, bipolar disorder (I, II, or NOS), schizophrenia or schizoaffective disorder, or anorexia nervosa.
* Current alcohol or drug dependence.
* Screening BDI ≥ 30 (severe depression).
* Known or suspected to have significant personality dysfunction that could, in the investigator's opinion, interfere with trial participation.
* Currently at risk of self-harm or harm to others, in the Sponsor's opinion, based on clinical interview.
* Currently a psychiatric inpatient; have been hospitalized for a psychiatric condition within the past year.
* Have ever been diagnosed with organic brain syndrome, mental retardation, or other cognitive dysfunction that could interfere with their capacity to participate in the study protocol.
* Body mass index ≥ 40 (in order to screen out individuals with Class III obesity who might be more prone to musculoskeletal injuries than individuals with a BMI < 40.0) or < 18.5 (in order to screen out individuals whose hormone levels may be impacted by their low weight).
* Resting blood pressure ≥ 160 systolic and/or 100 diastolic. Individuals currently being treated for high blood pressure and meeting these criteria are eligible.
* Receiving concurrent psychotherapy of any kind.
* Use of any psychotropic medications.
* Positive result on pregnancy test at Screening; plan to become pregnant during the course of the trial.
* Insufficient command of the English language (i.e., they cannot carry on a conversation with an interviewer in the English language or read associated text).

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2012-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Questionnaire | Weeks 0 (baseline) to 9 (post-intervention)
  The PSQ (Levenstein et al., 1993) is a self- report measure of cognitive and emotional reactions to perceived stressful situations. The questionnaire consists of four subscales assessing (1) worries, anxious concern for the future, feelings of desperation and frustration; (2) tension, exhaustion, and lack of relaxation; (3) positive feelings of challenge, joy, energy, and security; and (4) perceived environmental demands, such as lack of time, pressure, and overload.

SECONDARY OUTCOMES:
Feasibility | Weeks 0 (baseline) to 9 (post-intervention)
  Feasibility and acceptability of a yoga intervention for stress-induced eating. This interview, constructed by the PI, assesses participants' perceptions of ease of participation, program likeability, and perceived benefits of the yoga program. The interview consists of 16 open-ended questions.
Distress Tolerance | Weeks 0 (baseline) to 9 (post-intervention)
  The DTS (Simons & Gaher, 2005) is a 15-item self- report measure of physical and psychological distress tolerance.

OTHER OUTCOMES:
Depression Symptoms | Weeks 0 (baseline) to 9 (post-intervention)
  The BDI (Beck, Ward, Mendelson, Mock, & Erbaugh, 1961) is a widely used 21-item, self-report inventory that measures severity of depressive symptoms.
Anxiety Symptoms (BAI) | Weeks 0 (baseline) to 9 (post-intervention)
  The BAI (Beck, Epstein, Brown, & Steer, 1988) is a commonly used 21-item, self-report inventory designed to measure severity of anxiety symptoms.
Mindfulness | Weeks 0 (baseline) to 9 (post-intervention)
  Since yoga is a mindfulness based intervention, we will be looking at changes in mindfulness levels over the course of the intervention. ). The FFMQ (Baer et al., 2006) is a 39-item self-report measure of mindfulness components: observing, describing, acting with awareness, nonjudging of inner experience, and nonreactivity to inner experience.

CONTACTS AND LOCATIONS:
Overall Officials: Jasper Smits, Ph.D., Principal Investigator — Associate Professor
Locations (1):
- Southern Methodist University, Dallas, Texas, United States